CLINICAL TRIAL: NCT01785134
Title: Metabolic Effects of Different Surgical Methods to Treat Obesity
Brief Title: Effects of Different Surgical Methods to Treat Obesity
Acronym: DEOSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government); The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Erik Näslund, Professor, MD, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CT20110061; CT20110061 (Registry Identifier: Karolinska Clinical Trial Registration)
Record Dates: First submitted 2013-01-30; First posted 2013-02-07 (Estimated); Results first posted 2014-10-02 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2014-09

CONDITIONS: Obesity; Type 2 Diabetes; Insulin Sensitivity
Keywords: Obesity; Bariatric Surgery; Insulin Sensitivity
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Sham Comparator): Gastric bypass operation without omentectomy.
  Interventions: Procedure: Gastric bypass operation
- Omentectomy (Active Comparator): Gastric bypass operation in conjunction with removal of greater omentum
  Interventions: Procedure: Omentectomy; Procedure: Gastric bypass operation

INTERVENTIONS:
Procedure: Omentectomy
  Arms: Omentectomy
Procedure: Gastric bypass operation

SUMMARY:
Obese patients have an increased risk for developing severe metabolic disorders. This risk can only partly be reduced by weight reduction. The investigators have in a pilot study investigated if removal of abdominal fat (visceral) in addition to weight loss has additional beneficial effects on the metabolic profile and weight loss. This study aims to further investigate if removal of abdominal fat (major omentum) leads to beneficial metabolic effects.

ELIGIBILITY:
Inclusion Criteria:

Body mass index over 40 kg/m2

Body mass index over 35 kg/m2 with obesity associated co-morbidities such as type 2 diabetes and/or additional cardiovascular risk factors -

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, MD, PhD, Principal Investigator — Karolinska Institutet; Peter Arner, MD, PhD, Study Director — Karolinska Institutet; Johan Hoffstedt, MD, PhD, Study Chair — Karolinska Institutet
Locations (4):
- Sweden (4):
  - Södertälje Hospital, Södertälje, Stockholm County
  - Ersta Hospital, Stockholm, Stockholm County
  - Karolinska University Hospital Huddinge, Stockholm, Stockholm County
  - Danderyds Hospital, Stockholm, Stockholm County

REFERENCES:
- [Derived] van der Kolk BW, Muniandy M, Kaminska D, Alvarez M, Ko A, Miao Z, Valsesia A, Langin D, Vaittinen M, Paakkonen M, Jokinen R, Kaye S, Heinonen S, Virtanen KA, Andersson DP, Mannisto V, Saris WH, Astrup A, Ryden M, Blaak EE, Pajukanta P, Pihlajamaki J, Pietilainen KH. Differential Mitochondrial Gene Expression in Adipose Tissue Following Weight Loss Induced by Diet or Bariatric Surgery. J Clin Endocrinol Metab. 2021 Apr 23;106(5):1312-1324. doi: 10.1210/clinem/dgab072. PMID 33560372
- [Derived] Andersson DP, Thorell A, Lofgren P, Wiren M, Toft E, Qvisth V, Riserus U, Berglund L, Naslund E, Bringman S, Thorne A, Arner P, Hoffstedt J. Omentectomy in addition to gastric bypass surgery and influence on insulin sensitivity: a randomized double blind controlled trial. Clin Nutr. 2014 Dec;33(6):991-6. doi: 10.1016/j.clnu.2014.01.004. Epub 2014 Jan 12. PMID 24485000

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Gastric bypass operation without omentectomy.
  Gastric bypass operation
- Omentectomy: Gastric bypass operation in conjunction with removal of greater omentum
  Omentectomy
  Gastric bypass operation
Period: Overall Study
Arm/Group | Control | Omentectomy
Started | 41 | 40
Completed | 29 | 33
Not Completed | 12 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Omentectomy | Total
Number analyzed (Participants) | 41 | 40 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (9) | 43 (9) | 42 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 40 | 81
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 41 | 40 | 81

OUTCOME MEASURES:

1. Primary Outcome: Insulin Sensitivity at 2 Years
Description: Insulin sensitivity measured by hyperinsulinemic euglycemic clamp
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: glucose/kg body weight/min
Arm/Group | Control | Omentectomy
Number analyzed (Participants) | 29 | 33
glucose/kg body weight/min | 6.7 (1.6) | 6.6 (1.5)

2. Secondary Outcome: Body Composition at Two Years
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: % body fat
Arm/Group | Control | Omentectomy
Number analyzed (Participants) | 29 | 33
% body fat | 36 (8) | 38 (8)

3. Secondary Outcome: Blood Pressure at 2 Years
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: mm Hg systolic
Arm/Group | Control | Omentectomy
Number analyzed (Participants) | 29 | 33
mm Hg systolic | 123 (16) | 121 (23)

4. Secondary Outcome: Body Mass Index at 2 Years
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: Kg/meter squared
Arm/Group | Control | Omentectomy
Number analyzed (Participants) | 29 | 33
Kg/meter squared | 28.6 (4.6) | 28.9 (4.3)

5. Secondary Outcome: Blood Lipids
Time Frame: 2 years postoperative
Measure: Mean (Standard Deviation); unit: P-Cholesterol mmol/L
Arm/Group | Control | Omentectomy
Number analyzed (Participants) | 29 | 33
P-Cholesterol mmol/L | 4.0 (0.9) | 4.2 (0.8)

ADVERSE EVENTS:
Arm/Group | Control | Omentectomy
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40
Other Adverse Events (participants affected / at risk) | 0/41 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No